CLINICAL TRIAL: NCT05162885
Title: Effect of Sodium Alendronate Versus Sticky Bone as Socket Preservation Materials on the Final Implant Stability. A Randomized Clinical Trial
Brief Title: Effect of Sodium Alendronate on the Final Implant Stability.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hossam Abdallah Mohammed Ghazzaly, H.Ghazzaly, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: omfs335
Record Dates: First submitted 2021-12-07; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Anterior Labial Wall Defect
Keywords: Stability, Sodium Alendronate, Implant, Sticky bone
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- implant placement in defective Sockets preserved with alendronic acid sponge (Active Comparator): anesthesia according the site of implant placement were administered using mepivacaine HCl (2%) with levonordefrin 1:20 000 (Scandonest 2%; Septodont, Saint- Maur-des-Fossés, France). Injection to control pain and bleeding for hemostasis. Crestal incision with a full thickness mucoperiosteal flap was reflected .A pilot drill will be used to start the osteotomy preparation, then different drilling sizes will be used to attain the final drill size and the planed implant height and width according to Cone Beam CT. Implants were screwed directly into the osteotomy site, primarily the screwing was done mechanically by Fixture Mount Connection attached to the implant carrier.
  The created gap sutured passively to allow tension-free interrupted closure using 3-0 coated undyed braided polyglactin 910 suture material.
  Interventions: Procedure: Socket Preservation technique
- Implant placement in Defective sockets preserved with sticky bone (Active Comparator): anesthesia according the site of implant placement were administered using mepivacaine HCl (2%) with levonordefrin 1:20 000 (Scandonest 2%; Septodont, Saint- Maur-des-Fossés, France). Injection to control pain and bleeding for hemostasis. Crestal incision with a full thickness mucoperiosteal flap was reflected .A pilot drill will be used to start the osteotomy preparation, then different drilling sizes will be used to attain the final drill size and the planed implant height and width according to Cone Beam CT. Implants were screwed directly into the osteotomy site, primarily the screwing was done mechanically by Fixture Mount Connection attached to the implant carrier.
  The created gap sutured passively to allow tension-free interrupted closure using 3-0 coated undyed braided polyglactin 910 suture material.
  Interventions: Procedure: Socket Preservation technique

INTERVENTIONS:
Procedure: Socket Preservation technique — Implant placement after Socket preservation Technique with sodium alderonate versus sticky bone in salama&salama Class 3 labial wall defect
  Other Names: Implant in socket preserved with sodium alenderonate drug

SUMMARY:
evaluation of the final implant stability after its placement in sockets preserved with two different socket preservation materials

DETAILED DESCRIPTION:
compare the stability of implant placement using Osstell ISQ "resonance frequency analyzer", and marginal bone resorption and bone density around implant by X-ray analysis in different socket preservation techniques comparing sodium alendronate with the sticky bone graft technique

ELIGIBILITY:
Inclusion Criteria:

* Patients with seeking implant drive prosthesis after socket has been preserved by either technique.
* Patients with seeking implant drive prosthesis with Salama Class 3 defective sockets.
* Both genders males and females will be included.

Exclusion Criteria:

* General contraindications to implant surgery.
* Patient seeking immediate implant placement.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Active infection or severe inflammation in the area intended for implant placement.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly
* followed. Referred only for implant placement or unable to attend a 5-year follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 3-4 months after Dental implant placement
  Calculate the final implant stability of two groups using Osstell "resonance frequency analyzer"

SECONDARY OUTCOMES:
marginal bone | 3-4 months after Dental implant placement
  Evaluation of marginal bone resorption around implant in two groups using superimposition x-ray (CBCT) software analysis

OTHER OUTCOMES:
Bone Density | 3-4 months after Dental implant placement
  Evaluation of bone density around the placed implants using x-ray (CBCT) software analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam Abdallah Mohammed Ghazally, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No